CLINICAL TRIAL: NCT02548546
Title: Estimation of Biomechanical Aortic Wall Properties in Healthy and Aneurysmal Aortas Using Novel Imaging Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Houssam Farres, M.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-004151
Record Dates: First submitted 2015-08-26; First posted 2015-09-14 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Surveillance (Active Comparator): No Surgery with ECHO and ECG-gated MRA imaging.
  Interventions: Device: ECHO; Device: ECG-gated MRA
- Surgery-Open (Active Comparator): Open Surgery with ECHO and ECG-gated MRA imaging.
  Interventions: Device: ECHO; Device: ECG-gated MRA
- Surgery-EVAR (Active Comparator): EVAR with ECHO and ECG-gated MRA imaging.
  Interventions: Device: ECHO; Device: ECG-gated MRA

INTERVENTIONS:
Device: ECHO — Imaging
Device: ECG-gated MRA — Imaging

SUMMARY:
The primary aim of this study is to establish the practicality of using two novel imaging modalities for the assessment of biomechanical properties of the aorta.

DETAILED DESCRIPTION:
Patients with Abdominal Aortic Aneurysm, (AAA), will be identified within the vascular surgery practice. Those patients who meet standard indications for surgery including symptomatic AAA, size >5.0-5.5 cm, or rapidly enlarging >0.5 cm per 6 months will have standard pre-operative work-up which includes magnetic resonance angiogram (MRA) and Echocardiogram (ECHO). These pre-operative studies will be modified for the study patients to include electrocardiogram(ECG)-gating (coupled with MR angiogram) and 2-Dimensional speckle-tracking ultrasound of the abdominal aorta. Patients in the study will be followed for 1 year. Measurements will be analyzed for any relationship between aortic wall properties and clinical outcomes such as aneurysm growth, rupture risk or aortic dissection. This study will be comparing 3 groups of patients: no surgery (surveillance), open surgery, and endovascular aneurysm repair (EVAR).

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age with ability to provide informed consent.
* Patients with either symptomatic or asymptomatic AAA as defined by aortic diameter ≥ 1.5x normal diameter.
* Patients with non-aneurysmal aortas who require aortic contrast imaging or echocardiography for preoperative planning or other reason.

Exclusion Criteria:

* Patients with contraindication to IV contrast such as allergy or severe kidney dysfunction.
* Patients who do not require contrast imaging or echocardiogram as part of their care plan.
* Terminally ill patients, and patients with estimated life expectancy of ≤ 6 months.
* Patients unable to tolerate magnetic resonance imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
ECHO Imaging | Change from baseline in ECHO imaging measurements
  Imaging taken of the aneurysm, locating peak wall stress and measuring percent of strain per seconds.

SECONDARY OUTCOMES:
ECG-gated MRA Imaging | Change from baseline ECG-gated imaging measurements.
  The MRA imaging will be taken with the ECG-gating to synchronize the timing of the image acquisition with cardiac motion. This will allow for more accurate measurement of vessel diameter measured in mm (millimeters) and reported in percent change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Houssam Farres, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials